CLINICAL TRIAL: NCT01107535
Title: Observational Study of the Effectiveness of Synagis Immunoprophylaxis in Preterm Infants With High Risk of Severe Respiratory Syncytial Virus Infection
Brief Title: Effectiveness of Synagis (Palivizumab) Immunoprophylaxis in Preterm Infants With High Risk of Severe Respiratory Syncytial Virus (RSV) Infection
Acronym: INSPIRA
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: PMOS-PERU 07-01
Record Dates: First submitted 2010-02-20; First posted 2010-04-21 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Synagis (palivizumab) immunoprophylaxis; Respiratory syncytial virus infection; Preterm infants
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Palivizumab; Antibodies, Monoclonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Infants receiving Synagis (palivizumab) immunoprophylaxis: Infants born <= 32 weeks of gestation and are younger than 6 months of age, children with bronchopulmonary dysplasia who have received medical treatment in the last 6 months until the first year of life, and children 12 months or younger with hemodynamically significant acyanotic congenital heart disease (pulmonary hypertension or heart failure in treatment) prescribed Synagis (palivizumab) immunoprophylaxis according to the usual clinical practice.
  Interventions: Biological: Synagis (palivizumab), monoclonal antibody for passive immunoprophylaxis against severe RSV disease administered according to usual clinical practice.

INTERVENTIONS:
Biological: Synagis (palivizumab), monoclonal antibody for passive immunoprophylaxis against severe RSV disease administered according to usual clinical practice. — Synagis (palivizumab) administered according to usual clinical practice. After the enrollment visit, subjects will have monthly visits until they have received the complete Synagis immunization regimen of their hospital, then they will have 2 follow up visits, one of them 30 days after the fifth dose of Synagis and the other visit at one year of age.
  Other Names: palivizumab; Synagis

SUMMARY:
Published data by the Organización panamericana de la Salud shows that Peru's mortality rate from acute respiratory infections (ARI) in infants less than one year of life is second only to Haiti (14,150/100,000). Government data reports shows a marked increase of RSV infections in Peru. "Instituto Nacional de Salud" (Peru's National Institute of Health) reports between January 1st to February 26th 2006, 62% of their positive samples corresponded to RSV. Epidemiological data from Lima-Peru, demonstrates that there is no specific season for RSV infection although some data suggest an increase in RSV activity during cold months (May to September; INS data). Clinical studies show that giving five doses of Synagis (palivizumab) resulted in serum concentrations > 30 ug/mL for >20 weeks. The aim of this post-marketing observational study is to determine the RSV hospitalization rate in high-risk infants who received Synagis (palivizumab) through the Social Security Hospitals in the context of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Receiving Synagis (palivizumab) immunoprophylaxis during respiratory syncytial virus season, according to the usual clinical practice:
* Infants born < or = 32 weeks of gestation and are younger than 6 months of age at the beginning of the respiratory syncytial virus season.
* Children with bronchopulmonary dysplasia who have received medical treatment in the last 6 months, until the first year of life.
* Children 12 months or younger with hemodynamically significant acyanotic congenital heart disease (pulmonary hypertension or heart failure in treatment).

Exclusion Criteria:

* Major congenital malformation aside from congenital heart disease
* Chronic pulmonary disease other than bronchopulmonary dysplasia
* Active infections
* Contraindication to Synagis
* Receipt of another immunoglobulin preparation including but not restricted to polyclonal intravenous immunoglobulin, cytomegalovirus hyperimmunoglobulin (Cytogam), or respiratory syncytial virus hyperimmunoglobulin (Respigam).
* Any other condition that according deemed an obstacle for study conduction or representing an unacceptable risk by the participating investigator.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pre term neonates who received Synagis (palivizumab) according to the clinical practice. The study is implemented in 4 hospitals of Peru.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Guerra, MD, Study Director — Abbott
Locations (4):
- Peru (4):
  - Site Reference ID/Investigator# 27834, Arequipa
  - Site Reference ID/Investigator# 6059, Callao
  - Site Reference ID/Investigator# 27836, Lima
  - Site Reference ID/Investigator# 27835, Lima

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=23151&CFID

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Started | 82
Number of Participants Analyzed | 82
Completed | 77
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Number analyzed (Participants) | 82
Age Continuous [Mean (Standard Deviation); unit: days] — The mean age of participants at the first injection of study drug.
  days | 68 (63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 42
Region of Enrollment [Number; unit: participants]
  Peru | 82
Gestational age [Number; unit: participants] — Gestational age of participants.
  participants
    Gestational age less than 28 weeks | 22
    Gestational age >28 weeks and <32 weeks | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Hospital Admissions by Respiratory Syncytial Virus Infection
Description: The number of participants hospitalized for respiratory syncytial virus infection from the first dose of study drug up to the visit coinciding with the first birthday of the participant. An indirect immunofluorescence test (a laboratory technique used to detect the presence of viruses) was used to determine if hospitalized participants had respiratory syncytial virus infection.
Time Frame: First year of life (up to 12 months)
Population: Analysis included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Number analyzed (Participants) | 82
participants | 2

2. Secondary Outcome: Number of Hospital Admission Days (All Causes)
Description: The mean (average) number days participants were hospitalized.
Time Frame: Hospital admission to hospital discharge
Population: Analysis included all participants who were hospitalized during the study. This includes 2 participants hospitalized due to respiratory syncytial virus infection and 8 participants hospitalized for other respiratory diseases.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Number analyzed (Participants) | 10
days | 18.4 (29.7)

3. Secondary Outcome: Number of Intensive Care Unit Days During the Hospital Admissions by Respiratory Syncytial Virus Infection
Description: The number of days spent in a hospital intensive care unit (ICU) are summarized for those participants requiring that type of care. An indirect immunofluorescence test (a laboratory technique used to detect the presence of viruses) was used to determine if hospitalized participants had respiratory syncytial virus infection.
Time Frame: Hospital admission to hospital discharge
Population: Two participants with a total of 3 intensive care unit stays were analyzed. One participant was negative for respiratory syncytial virus during their first stay in the intensive care unit and was positive for respiratory syncytial virus at their second stay.
Measure: Number; unit: days
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Number analyzed (Participants) | 2
days
  ICU stay length (n=1, RSV negative) | 5
  ICU stay length (n=1, Stay #1 of 2, RSV negative) | 10
  ICU stay length (n=1, Stay #2 of 2, RSV positive) | 106

4. Secondary Outcome: Number of Ventilation Support Days (Supplemental Oxygen and Mechanical Ventilation) During the Hospital Admission
Description: The mean (average) number of days participants required supplemental oxygen during any hospital stay and the mean number of days participants required mechanical ventilation while in the intensive care unit.
Time Frame: Hospital admission to hospital discharge
Population: Analysis of supplemental oxygen included participants with any hospital stay during the study (n=10) and analysis of mechanical ventilation included the subgroup of participants with intensive care unit stays during the study (n=2).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Number analyzed (Participants) | 10
days
  Supplemental oxygen (n=10) | 17 (32)
  Mechanical ventilation (n=2) | 36.7 (49)

5. Secondary Outcome: Number of Serious Adverse Events
Description: The number participants experiencing a serious adverse event. For additional information see the Reported Adverse Events section.
Time Frame: Enrollment until 100 days after the last Synagis (palivizumab) dose
Population: Analysis included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Number analyzed (Participants) | 82
participants | 11

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the study observation period until 100 days after the last dose of Synagis. Participants were followed for an average of 12.4 months.
Arm/Group | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis
Serious Adverse Events (participants affected / at risk) | 11/82
Other Adverse Events (participants affected / at risk) | 17/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis (N=82)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory syncytial virus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retinopathy of immaturity (Eye disorders) | 1 (1)
Sudden infant death syndrome (General disorders) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants Receiving Synagis (Palivizumab) Immunoprophylaxis (N=82)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.